CLINICAL TRIAL: NCT01598285
Title: A Combined Genome-Wide Association Study (GWAS) and microRNA (miRNA) Profiling Approach for the Identification of Bevacizumab Response Predictors in Metastatic Breast Cancer
Brief Title: A Combined GWAS and miRNA for the Identification of Bevacizumab Response Predictors in Metastatic Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Due to the low rate of recruitment.
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Hoffmann-La Roche (Industry); Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: GEICAM/2011-07; GEICAM/2011-07 (Other: GEICAM/2011-07)
Record Dates: First submitted 2012-04-20; First posted 2012-05-15 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer Invasive Nos
Keywords: Genome-Wide; GWAS; microRNA; miRNA; Bevacizumab Response Predictors; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
GEI-BEV-2011-01 is an Observational multicenter study. The study, involving 200 (100 non-responders and 100 best responders) metastatic breast cancer patients, will search for specific genetic variants (SNPs) and miRNA signatures associated with bevacizumab response. Only patients suffering from metastatic (disseminated at the time of diagnosis) breast cancer, treated with bevacizumab, will be included.

1. -To identify genetic variants as bevacizumab response predictors in metastatic breast cancer
2. To identify miRNA signatures in whole blood as bevacizumab response predictors in metastatic breast cancer patients.

The main endpoint will be progression-free survival (PFS)

The duration of the study will be approximately 18 months

DETAILED DESCRIPTION:
In certain solid neoplasias, antiangiogenic therapies improve response rates and time to progression. However, treatment with antiangiogenic drugs do not improve patient´s overall survival, in addition to being quite toxic and expensive. It is therefore critical to identify reliable predictive factors for drug efficacy and potential toxicity. Pharmacogenomics and pharmacogenetics are emerging as important tools in the optimization of different therapeutic strategies against cancer. Thus, gene expression profiling and genome-wide association studies (GWAS) offer the promise to more effectively tailor individual cancer treatments by identifying new biomarkers for clinical efficacy. They likely represent a real progress in our understanding of cancer as a complex process and an improvement in patient management and treatment. This grant proposal is aimed at: i) identify genetic variants (SNPs) responsible for the different bevacizumab treatment response observed in metastatic breast cancer patients and ii) determine specific blood microRNA (miRNA) signatures associated with the bevacizumab response The reference endpoint for patient selection will be progression free survival (PFS). To increase the statistical significance of the study, patients will be categorized in two groups: non-responders (PFS<12 weeks) and best responders (PFS>52 weeks). Blood samples will be drawn prospectively from selected patients, they will be processed to obtain purified total DNA and RNA and, finally, they will be analyzed by next-gen GWAS and miRNA profiling, respectively. DNA samples will be hybridized to ultrahigh density Omni microarrays, containing 2.5 million genetic variants while RNA samples will be hybridized to Affymetrix microarrays containing an up-to-date collection of human miRNA sequences (miRBase v15, 1105 human miRNA probes). Standard computational analysis of both sets of microarray data will performed and the results will be correlated with the main endpoint of the study (PFS).

ELIGIBILITY:
Inclusion Criteria:

* patients with breast cancer, at a disseminated stage
* patients treated with bevacizumab in combination with weekly paclitaxel as first line chemotherapy and who have progressed
* alive patients authorizing the extraction and analysis of their biological samples.

Exclusion Criteria:

* patients with a second neoplasia
* deceased patients
* patients who have not agreed to participate in the study
* HER2 positive patients
* patients with CNS metastases when first treated with bevacizumab in combination with paclitaxel
* patients with local-regional recurrence only and
* patients with status NED (resected metastases)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from metastatic (disseminated at the time of diagnosis) breast cancer, treated with bevacizumab.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-04-18 (Actual); Primary Completion 2013-04-10 (Actual); Study Completion 2013-04-10 (Actual)

PRIMARY OUTCOMES:
Genome-Wide Association Study (GWAS) and microRNA (miRNA) profiling for identification of genetic variants and blood miRNA signatures predictors of bevacizumab response. | 18 months
  Genome-Wide Association Study (GWAS) and microRNA profiling will be performed from DNA and microRNA obtained from blood samples of metastatic breast cancer patients treated with Bevacizumab. Next-generation microarray thecnologies will be performed. Patients will be categorized in two groups: non-responders and best responders. Results of standard computational analysis of microarrays will be correlated with progression free survival data for identification of genetic variants and microRNA signatures predictors of Bevacizumab response

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Clínico Universitario Virgen de la Victoria
Locations (1):
- Hospital Clínico Universitario Virgen de la Victoria, Málaga, Spain

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org